CLINICAL TRIAL: NCT01516177
Title: An Observational Study to Assess the Prevalence of a Tolerance Signature in Renal Transplant Recipients (ITN524ST/CTOT-12)
Brief Title: Associating Renal Transplantation With the ITN Signature of Tolerance
Acronym: ARTIST
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Immune Tolerance Network (ITN) (Network); Clinical Trials in Organ Transplantation (Network)
Responsible Party: Sponsor
Other Study IDs: DAIT ITN524ST/CTOT-12
Record Dates: First submitted 2012-01-19; First posted 2012-01-24 (Estimated); Last update posted 2016-12-20 (Estimated); Status verified 2016-12

CONDITIONS: Kidney Transplantation
Keywords: Kidney Transplantation; kidney transplant; renal transplant; immunosuppression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood Isolation PBMC isolated RNA specimens
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Renal Transplant Recipients: Subjects who received a kidney transplant within the past 1 to 5 years

SUMMARY:
This is an observational study for people who have received a kidney transplant within the past 1 to 5 years. Researchers in this study are looking for a certain pattern of genes and cells in the blood that has been found in a group of rare transplant patients who do not need immunosuppression. The study goal is to find out how common this pattern is in transplant patients, as a first step in determining if it can be used to personalize anti-rejection drug regimens better.

DETAILED DESCRIPTION:
Following surgery, kidney transplant patients must take medications in order to prevent rejection of their transplanted organ. These medications can be very effective. Called immunosuppressive drugs, they work by reducing the activity of the immune system. Because of this, however, they can also have serious side effects, including increased risks of serious infections and certain types of cancer.

The ITN Registry of Tolerant Kidney Transplant Recipients recently identified a rare group of people whose immune system has accepted their transplant without continued use of immunosuppressive drugs. Researchers have found that these patients have a unique pattern of cells and genes expressed in their blood compared to other transplant patients.

The ARTIST study will ask the questions "Are there other transplant patients who show this pattern?" and "If so, how often?"

The goal is to find out if there are other transplant patients who are taking immunosuppression who also show this pattern of genes. If there are others, then this pattern may one day be useful in identifying transplant patients who could reduce the dose of immunosuppression they need without fear of rejection.

Researchers are seeking adults who have received a kidney transplant within the past 1 to 5 years. Participants will be asked to attend 3 short appointments with study doctors over a period of 2 years. At these visits, doctors will request demographic and clinical information, relevant medical histories and blood and urine samples. Participants will be compensated for their time.

It is important to note that this is an observational study only. Other than receiving consultations and advice from the transplant team, there is no direct medical benefit to participating. However, by participating, patients may play an active part in helping doctors learn to control kidney transplant rejection more effectively, with fewer drugs.

ELIGIBILITY:
Inclusion Criteria:

* Received first kidney transplant from a living or deceased donor.
* Kidney transplanted between 1 and 5 years ago.
* Calculated GFR of greater than or equal to 45 mL/min/1.73 m2 within last 6 months
* Ability to understand and provide informed consent.

Exclusion Criteria:

* History of steroid-resistant acute rejection
* History of two or more episodes of acute rejection
* Any acute rejection in the past year
* Current malignancy
* Transplant of another organ
* AIDS according to the CDC definition of AIDS.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include 250 participants who are determined to be eligible for further follow-up based on the eligibility criteria.
  Among those eligible for further follow-up
  * at least 25 participants will be renal transplant recipients who received induction therapy with Campath, and
  * at least 25 participants will be renal transplant recipients who are receiving sirolimus or everolimus at time of enrollment and who have not received calcineurin inhibitors for at least 30 days prior to enrollment
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2010-09; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
The presence of at least one time point of the previously identified renal transplant tolerance signature. | 2 years

SECONDARY OUTCOMES:
Time course of potential changes in the previously identified renal transplant tolerance signature in individual participants. | 2 years
Expression levels for a wide variety of genes measured by large-scale microarray or by PCR assessments | 2 years
Flow-cytometric measurements of cell populations distinguished by cell-surface phenotype | 2 years
Selected clinical events and laboratory parameters to assess hematologic and renal function | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Anil Chandraker, MD, Study Chair — Brigham and Women's Hospital; Kenneth Newell, MD, PhD, Study Chair — Emory University; Laurence Turka, MD, Study Chair — Beth Israel Deaconess Medical Center
Locations (8):
- United States (8):
  - University of Alabama Birmingham, Birmingham, Alabama
  - University of California San Francisco, San Francisco, California
  - Emory University, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Mount Sinai School of Medicine, New York, New York
  - The Cleveland Clinic Foundation, Cleveland, Ohio

REFERENCES:
- [Background] Newell KA, Asare A, Kirk AD, Gisler TD, Bourcier K, Suthanthiran M, Burlingham WJ, Marks WH, Sanz I, Lechler RI, Hernandez-Fuentes MP, Turka LA, Seyfert-Margolis VL; Immune Tolerance Network ST507 Study Group. Identification of a B cell signature associated with renal transplant tolerance in humans. J Clin Invest. 2010 Jun;120(6):1836-47. doi: 10.1172/JCI39933. Epub 2010 May 24. PMID 20501946
- See also: National Institute of Allergy and Infectious Diseases (NIAID) website — https://www.niaid.nih.gov/
- See also: Immune Tolerance Network website — http://www.immunetolerance.org
- See also: Clinical Trials in Organ Transplantation website — https://www.ctotstudies.org/